CLINICAL TRIAL: NCT00200395
Title: Phase II Study of OSI-774 (Erlotinib, Tarceva) in Elderly Patients With Advanced Stage or Inoperable Non Small Cell Lung Cancer (NSCLC)
Brief Title: OSI-774 (Erlotinib, Tarceva) in Elderly Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-01-019
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OSI-774 (Tarceva) (Experimental): Oral treatment with OSI-774 (Tarceva) will be given as a 150 mg tablets daily for 14 days. On day 15 and if there are no adverse effects the dose will be increased to 200 mg.
  Interventions: Drug: Tarceva

INTERVENTIONS:
Drug: Tarceva — OSI-774 will be supplied as 25 mg (non -film coated) 100 and 150 mg (film coated) tablets in separate bottles, containing 30 tablets respectively.
  Other Names: OSI-774; Erlotinib

SUMMARY:
The purpose of this research study is to determine if OSI-774 (Tarceva) is effective in the treatment of non-small cell lung cancer and to further study its side effects. The investigators would also like to estimate disease-related symptom improvement rates using a questionnaire.

DETAILED DESCRIPTION:
In recent years, it has been shown that the degree of improvement achievable with chemotherapy has plateaued with the use of chemotherapy doublets. The presence of co-morbid conditions and poor performance status may preclude the use of chemotherapy in many elderly patients, which even in the medically fit, has modest benefits. The advent of targeted cancer therapy with the discovery of tyrosine kinases as mediators of tumor growth, with its limited toxicity profile, offers a promising approach to the treatment of NSCLC, in particular to the elderly subset of patients. The encouraging results from the other trials provide a strong rationale to evaluate an oral EGFR-tyrosine kinase inhibitor OSI-774 in patients with advanced and inoperable NSCLC over the age of 70. In vitro and clinical data suggest a dose- dependent response with Tarceva (Genentech, data on file).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have confirmed non-small cell lung cancer. Age > 65 years Patients must have adequate organ and marrow function

Exclusion Criteria:

* Patients who have had prior chemotherapy will be excluded. Patients may not be receiving any other investigational agents.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-07-02 (Actual); Primary Completion 2007-01-12 (Actual); Study Completion 2007-01-12 (Actual)

PRIMARY OUTCOMES:
Rate of Response | 1-3 years
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date the recurrent or progressive disease is documented.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v2.0 | 1-3 years
Changes in Quality of Life (QOL): questionnaire | through study completion, an average of 3 years
  This will involve participant response to a seven-item lung cancer subscale of Functional Assessment of Cancer Therapy-Lung (FACT-L) questionnaire.
Rate of Progression free survival | 1-3 years
  Progression free survival is defined as the duration of time from start of treatment to time of progression.
Duration of stable disease | 1-3 years
  Stable disease is measured from the start of the treatment until the criteris for progression are met., taking as reference the smallest measurements recorded since the treatment started.
Overall Rate of Survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi Rajdev, M.D., Study Chair — Montefiore Medical Center
Locations (4):
- United States (4):
  - Beth Israel Medical Center, New York, New York
  - New York University, New York, New York
  - Albert Einstein Cancer Center, The Bronx, New York
  - Montefiore Medical Center-, The Bronx, New York